CLINICAL TRIAL: NCT04750603
Title: Fluticasone Furate/Vilaterol in Exercising Asthmatic Adolescents: a Randomized and Open Label Trial
Brief Title: Effect of Fluticasone Furoate/Vilanterol on EIA in Adolescents
Acronym: EIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, l_bentur, Prof. Lea Bentur, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMB-107-18
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Asthma in Children
MeSH Terms: interventions — fluticasone furoate; Albuterol

STUDY DESIGN:
Intervention Model Description: First phase: Randomized, double blind, double dummy. Second phase: open label
Who Masked: Participant, Investigator
Masking Description: Medications and placebos were provided by the hospital pharmacy and medications were given by the nurse. Randomization was generated by computer, independently of trial staff as described (Salbutamol inhaler + Ellipta placebo or FF/VI + placebo Salbutamol inhaler). Technicians performing the ECT, investigators and patients were blinded to treatment choice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salbutamol (Placebo Comparator): Salbutamol (Salbutrim, Trima) inhaler (400 µg) via spacer + Relvar® Ellipta placebo
  Interventions: Drug: Salbutamol
- FF/VI (Active Comparator): Placebo Salbutamol inhaler + Relvar® Ellipta (92/22 µg, GSK, UK)
  Interventions: Drug: Fluticasone furoate (FF)/Vilanterol (VI)

INTERVENTIONS:
Drug: Fluticasone furoate (FF)/Vilanterol (VI) — Patients with a positive exercise challenge test were allocated to a single administration of salbutamol (400 µg) and 22 to FF/VI (92/22 µg) in a double blind, double dummy method to assess the short-term effect on exercise induced complaints
  Other Names: Relvar®
  Arms: FF/VI
Drug: Salbutamol — Patients with a positive exercise challenge test were allocated to a single administration of salbutamol (400 µg) and 22 to FF/VI (92/22 µg) in a double blind, double dummy method to assess the short-term effect on exercise induced complaints.
  Other Names: Salbutrim
  Arms: Salbutamol

SUMMARY:
Exercise induced asthma (EIA) is common in adolescents. (Fluticasone furoate (FF)/Vilanterol (VI)) is a once daily inhaler with bronchodilator effect lasting 24 hours. Our objective was to investigate the short and long-term effects of FF/VI on EIA in adolescents. Adolescent asthmatics were referred for evaluation of EIA. Patients with a positive exercise challenge test, were allocated to a single administration of salbutamol and 22 to FF/VI in a double blind, double dummy method to assess the short-term effect on EIA. Then they received FF/VI for 30-60 days and were reassessed by a repeat exercise test 24-hours after the last dose.

DETAILED DESCRIPTION:
Exercise induced asthma (EIA) is common in adolescents. Relvar® (Fluticasone furoate (FF)/Vilanterol (VI)) is a once daily inhaler with bronchodilator effect lasting 24 hours. Our objective was to investigate the short and long-term effects of FF/VI on EIA in adolescents. Ninety-three adolescent asthmatics aged 12-18 years were referred for evaluation of EIA. 44 patients had a positive exercise challenge test (ECT), 22 (22/44) were allocated to a single administration of salbutamol (400 µg) and 22 to FF/VI (92/22 µg) in a double blind, double dummy method to assess the short-term effect on EIA. Then they received FF/VI for 30-60 days and were reassessed by a repeat ECT 24-hours after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent asthmatics aged 12-18 years
* Symptoms of shortness of breath on exercise and asthmatics before entry to military service
* Referral for evaluation of exercise challenge test

Exclusion Criteria:

* Baseline FEV1<65% before exercise test
* Acute illness
* History of intolerance to beta agonists
* Use of the following medications prior to the study was restricted: inhaled corticosteroids or Montelukast (2 weeks), systemic steroids (2 months) and bronchodilators (24 hours)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Long term effect of FF/VI | 30-60 days
  Exercise challenge test following FF/VI treatment

SECONDARY OUTCOMES:
Short term effect of FF/VI | 15 minutes
  Effect of FF/VI on post exercise change in pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Rambam
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be available.